CLINICAL TRIAL: NCT04118439
Title: Effectiveness of an Exercise Program Combined With Action Observation and Motor Imagery in Patients With Chronic Shoulder Pain in Primary Care. A Controlled Clinical Trial
Brief Title: Effectiveness of Action Observation and Motor Imagery Intervention Plus Exercise for Chronic Painful Shoulder in Primary Care
Acronym: OPTIMIST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Raúl Ferrer-Peña, Professor and Researcher, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI-4001
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Shoulder Pain
Keywords: Motor Imaginery; Shoulder Pain; Chronic Pain
MeSH Terms: conditions — Shoulder Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imaginery (Experimental): Patients allocated in this arm will recieve a training on the first day after recruitment on a motor imaginery task and will be asked to do the task every day during 30 days until they start the usual care. Then after the physical therapy treatment with a pragmatic perspective will be meassured just inthe last session, after 1 month an.d after 3 moths of the treatment for the follow up
  Interventions: Other: Motor Imaginery and Action Observation
- Control Group (No Intervention): Patients allocated in this arm will be meassured at the start, again after 30 days and at the end of the physical therapy usual care with a pragmatic perspective. Then will be meassured again after 1 and 3 months.

INTERVENTIONS:
Other: Motor Imaginery and Action Observation — A set of tasks done with the shoulder, first with an Action Observation perspective and then asked to perform this tasks with motor imaginery
  Arms: Motor Imaginery

SUMMARY:
Objective: to evaluate the effectiveness of an action observation program (OA) and motor imagery (MI) -integrated into routine physiotherapy practice- to reduce disability associated with chronic shoulder pain in primary care, after 8 weeks of intervention and with follow-ups at 3 and 6 months with blind evaluation of the response variable. Design: randomized controlled clinical trial. Population: Patients with chronic shoulder pain diagnosed and referred by their family doctors to the physiotherapy service will be included. Intervention: Group: experimental: MI+OA+ multicomponent exercises or control group: multicomponent exercises. 100 patients (50 per group) will be included. Variables: sociodemographic and clinical variables will be collected.

Primary variable: Disability related to pain in the shoulder region; Secondary variables: Intensity of perceived pain, Shoulder Joint Range of Motion, Hand and shoulder strength, Fear of movement, Catastrophizing in the face of pain, Quality of life of patients, Global Perception of Change, and adherence to exercise. Statistical analysis: Descriptive. Main effectiveness analysis by intention to treat comparing the difference between groups in the average disability for the different intervention times.

Multivariate analysis considers the influence of psychological variables on pain and on the therapeutic response. An analysis segmented by sex will be carried out, and the influence of psychological variables on pain and on the therapeutic response will be analyzed.

DETAILED DESCRIPTION:
The aim of this project is to investigate a new conservative therapeutic approach for patients with chronic shoulder pain, a highly prevalent condition in primary care, and with a significant percentage of patients experiencing persistent pain. The proposed intervention combines Action Observation (AO) and Motor Imagery (MI) techniques with the usual based on exercises, with the aim of enhancing its effects by reducing disability, improving adherence to treatment and reducing the impact of pain on recovery. Although these techniques have been little explored in shoulder rehabilitation, they have scientific evidence in other areas of neuromusculoskeletal rehabilitation.

The study will be carried out in primary care, with the aim of improving the quality of the treatments available in these centers. The intervention will facilitate compliance with home treatment guidelines, which will shorten recovery times and sick leave, thus optimizing access to rehabilitation services for new patients.

A key component of the project will be the dissemination of results, both in the scientific community and in society. In addition to scientific publications and conference presentations, various dissemination strategies will be implemented: 1) Social networks social networks: Publication of summaries, graphics and explanatory videos about the project and its findings. 2) Teaching materials and practical guides : Development of resources aimed specifically at primary care physiotherapists to facilitate the implementation of the techniques in clinical practice. 3) Public awareness: Dissemination of information about chronic shoulder pain and advances in its treatment, through articles, press releases and interviews in specialized and general media.

This comprehensive approach will not only scientifically validate the intervention, but also transfer knowledge to health professionals and society, promoting a more accessible and effective treatment for patients with chronic shoulder pain

.

ELIGIBILITY:
Inclusion Criteria:

1. who have been diagnosed and referred by the family physician to physiotherapy units in primary care by a process of muscular origin in the shoulder region,
2. who have not received physiotherapy treatment by the same process in the last 6 months.

Exclusion Criteria:

1. suffer from systemic diseases such as rheumatoid arthritis, fibromyalgia, diagnosed neurological disease, lupus erythematosus, or cancer.
2. History of shoulder surgery,
3. patients with psychiatric pathologies or personality disorders;
4. patients with severe mobility limitation compatible with the diagnosis of frozen shoulder, 5) patients diagnosed with type II diabetes,

6) patients with little knowledge of Spanish language spoken or written and 7) reproduction of symptoms during active movements of the cervical spine or during palpation of the cervical or thoracic region.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Previous the intervention
  Pain Intensity with Visual Analogue Scale (range: 0-10). Higher scores mean more intensity
Change in Pain Intensity | At 30 days from the begining finishing the intervention
  Pain Intensity with Visual Analogue Scale (range: 0-10). Higher scores mean more intensity
Change in Pain Intensity | At the end of the usual care period of 4 weeks
  Pain Intensity with Visual Analogue Scale (range: 0-10). Higher scores mean more intensity
Change in Pain Intensity | Up to 12 weeks
  Pain Intensity with Visual Analogue Scale (range: 0-10). Higher scores mean more intensity

SECONDARY OUTCOMES:
Shoulder Disability: SPADI questionnaire | Previous the intervention
  Shoulder Disability with SPADI questionnaire (range: 0-100). Higher scores mean more disability
Change in Shoulder Disability | Up to 12 weeks
  Shoulder Disability with SPADI questionnaire (range: 0-100). Higher scores mean more disability
Health Related Quality of Live | Previous the intervention
  Health Related Quality of Live with EuroQoL-5D-5L (range 11111 - 55555). Higher scores mean worst Quality of Life
Change in Health Related Quality of Live | Up to 12 weeks
  Health Related Quality of Live with EuroQoL-5D-5L (range 11111 - 55555). Higher scores mean worst Quality of Life
Pain Catastrophizing | Previous the intervention
  Pain Catastrophizing with Pain Catastrophizing Scale (range 0-52). Higher scores mean more catastrophizing
Change in Pain Catastrophizing | Up to 12 weeks
  Pain Catastrophizing with Pain Catastrophizing Scale (range 0-52). Higher scores mean more Catastrophizing
Pain Severity | Previous the intervention
  Pain Severity with Graded Chonic Pain Scale (rango 0-70). Higher scores mean more severity
Change in Pain Severity | Up to 12 weeks
  Pain Severity with Graded Chonic Pain Scale (rango 0-70). Higher scores mean more severity
Change Perception | At 12 weeks from the end of the intervention
  Change Perception with Global Rating of Change Scale (range -5 to + 5). - 5 means worst than before and +5 means Completely recovered

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luime JJ, Koes BW, Hendriksen IJ, Burdorf A, Verhagen AP, Miedema HS, Verhaar JA. Prevalence and incidence of shoulder pain in the general population; a systematic review. Scand J Rheumatol. 2004;33(2):73-81. doi: 10.1080/03009740310004667. PMID 15163107
- [Background] Tinazzi M, Fiaschi A, Rosso T, Faccioli F, Grosslercher J, Aglioti SM. Neuroplastic changes related to pain occur at multiple levels of the human somatosensory system: A somatosensory-evoked potentials study in patients with cervical radicular pain. J Neurosci. 2000 Dec 15;20(24):9277-83. doi: 10.1523/JNEUROSCI.20-24-09277.2000. PMID 11125006
- [Background] Eaves DL, Riach M, Holmes PS, Wright DJ. Motor Imagery during Action Observation: A Brief Review of Evidence, Theory and Future Research Opportunities. Front Neurosci. 2016 Nov 21;10:514. doi: 10.3389/fnins.2016.00514. eCollection 2016. PMID 27917103